CLINICAL TRIAL: NCT04328922
Title: Fecal Microbial Transplantation for the Optimization of Vedolizumab Treatment in Patients With Crohn's Disease
Brief Title: Fecal Microbial Transplantation and Vedolizumab Treatment of Crohn's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Head of R&D development, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-16-NH-0123-CTIL
Record Dates: First submitted 2019-02-08; First posted 2020-04-01 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Crohn Disease; Microbial Substitution
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: A randomized double blinded controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients, treating physician and study investigators will be blinded to the treatment intervention (FMT/ placebo).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fecal microbial transplantation (Active Comparator): FMT capsules fecal capsules on two consecutive days (total of 30 capsules) within a week prior to first vedolizumab infusion. Patients who will be allocated to this treatment arm will be matched to donors according to their CMV status (past exposure - CMV positive donors will be used for CMV positive patients, and CMV negative donors will be used for CMV negative patients).
  Interventions: Other: Fecal microbial transplantation
- Placebo (Placebo Comparator): Placebo capsules placebo capsules- on two consecutive days (total of 30 capsules) within a week prior to first vedolizumab infusion. Patients who will be allocated to this treatment arm will receive placebo capsules.
  Interventions: Other: Placebo capsuls

INTERVENTIONS:
Other: Fecal microbial transplantation — Capsules of fecal matter solution (feces from healthy donor, glycerol and saline solution)/
  Arms: Fecal microbial transplantation
Other: Placebo capsuls — capsules of glycerol and saline (placebo).
  Arms: Placebo

SUMMARY:
The investigators postulate that by determining a patient's baseline microbiome and manipulating it through fecal microbial transplantation (FMT) may improve response rates to vedolizumab in Crohn's disease (CD) patients.

Primary objective: To determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is safe and results in higher remission rates in CD patients.

Study design: A randomized double blinded controlled clinical trial. Study population:CD patients 18-65 YO, men and women, with mild-moderately active disease determined by the Harvey-Bradshaw index (HBI) of 5≤HBI≤15, who were found eligible to commence treatment with vedolizumab.

Study procedure: Study participants will receive FMT within a week prior to first vedolizumab infusion.

All patients will be followed for 46 weeks in 8 visits at the IBD clinic in the GI department of the Tel Aviv Medical Center.

DETAILED DESCRIPTION:
Study design: A randomized double blinded controlled clinical trial.

Study population:

CD patients 18-65 YO, men and women, with mild-moderately active disease determined by the Harvey-Bradshaw index (HBI) of 5≤HBI≤15, who were found eligible to commence treatment with vedolizumab (screened for tuberculosis and hepatitis B and without an active infection or an abscess) will be enrolled in the study.

Follow-up: All patients will be followed by physician assessment, sample collection, anthropometric measurements and questionnaires during the scheduled visits at weeks 2, 6, 14, 22, and at week 46, on which they will undergo a colonoscopic examination as part of their regular clinical followup.

Side effects (SE): will be monitored by phone, 3 days post intervention and at vedolizumab infusion visits at weeks 2 and 6. Also, patients will receive direct contact details of both the study coordinator and the study PI.

ELIGIBILITY:
Inclusion Criteria:

1. Mild-moderately active disease determined by the Harvey-Bradshaw index (HBI) of 5≤HBI≤15
2. Found eligible to commence treatment with vedolizumab (screened for tuberculosis and hepatitis B and without an active infection or an abscess)

Exclusion Criteria:

1. CD patients in remission (HBI<5) or with sever disease (HBI>16)
2. Patients with a stoma
3. Hospitalized patients
4. Patients with an active intestinal infection- positive stool culture or Clostridium difficile infection
5. Severe disease - malignant disease, hepatic failure, renal failure, cardiovascular, metabolic, neurological disease
6. Pregnant/lactating women
7. Inability to sign an informed consent
8. Inability to complete the study protocol
9. An ongoing or planned antibiotics therapy
10. Severe food allergies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-07-03 (Actual); Primary Completion 2022-04 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
safety of FMT pre vedolizumab treatment in CD patients | week 14
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is safe.
  safety of FMT will be measured by disease exacerbations, hospitalizations and surgery rate in treatment versus placebo group.
safety of FMT pre vedolizumab treatment in CD patients: measured by disease exacerbations, hospitalizations and surgery rate in treatment versus placebo group | week 46
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is safe.
  safety of FMT will be measured by disease exacerbations, hospitalizations and surgery rate in treatment versus placebo group.
efficacy of FMT pre vedolizumab treatment in CD patients that results in higher remission rate | week 14
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is efficient and results in higher remission rates in CD patients.
  Remission rate will be measured by clinical remission rate HBI ≤5 at week 14
efficacy of FMT pre vedolizumab treatment in CD patients that results in higher remission rate | week 46
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is efficient and results in higher remission rates in CD patients.
  Remission rate will be measured by clinical remission rate HBI ≤5 at week 46

SECONDARY OUTCOMES:
efficacy of FMT pre vedolizumab treatment in CD patients that results in clinical response rate | week 14
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is efficient and results in clinical response rate (reduction in HBI≥3 )
efficacy of FMT pre vedolizumab treatment in CD patients that results in clinical response rate | week 22
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is efficient and results in reduction in HBI≥3
efficacy of FMT pre vedolizumab treatment in CD patients that results in clinical response rate | week 46
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is efficient and results in reduction in HBI≥3
efficacy of FMT pre vedolizumab treatment in CD patients that results in endoscopic response | week 46
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is efficient and results in endoscopic response that will be defined as a decrease of ≥50% in SES-CD score / improvement in Rutgeerts score ≥1, compared to baseline colonoscopy
efficacy of FMT pre vedolizumab treatment in CD patients that results in endoscopic remission | week 46
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is efficient and results in Endoscopic remission at week 46 will be defined as SES-CD ≤2 or Rutgeerts score ≤1 , compared to baseline colonoscopy
efficacy of FMT pre vedolizumab treatment in CD patients that results in histological healing | week 46
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is efficient and results in histological healing compared to week 0
efficacy of FMT pre vedolizumab treatment in CD patients that results in biological remission | week 14
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is efficient and results in biological remission measured as fecal calprotectin<150mg/kg and CRP<5mg/L
efficacy of FMT pre vedolizumab treatment in CD patients that results in biological remission | week 22
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is efficient and results in biological remission measured as fecal calprotectin<150mg/kg and CRP<5mg/L
efficacy of FMT pre vedolizumab treatment in CD patients that results in biological remission | week 46
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is efficient and results in biological remission measured as fecal calprotectin<150mg/kg and CRP<5mg/L
safety of FMT pre vedolizumab treatment in CD patients that results in low adverse events rate | week 46
  determine whether manipulation of gut microbiome by FMT pre vedolizumab treatment is safe and results in lower adverse events rate of intervention versus placebo

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Department of Gastroentherology, Tel Aviv
  - Dep. of Gastroenterology, Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No